CLINICAL TRIAL: NCT04496089
Title: Open-label Phase I of 89Zr-girentuximab (89Zr-TLX250) to Assess the Safety, Biodistribution, Pharmacokinetics and Sensitivity/Specificity of PET/CT Images in Patients With Suspected Renal Cell Carcinoma Including Clear Cell Renal Cell Carcinoma (ZIRDAC-JP Study)
Brief Title: Evaluation of Safety, Biodistibution and Sensitivity/Specificity of PET/CT Imaging With 89Zr-TLX250 in Subjects With RCC
Acronym: ZIRDAC-JP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 89Zr-TLX250-004
Record Dates: First submitted 2020-07-14; First posted 2020-08-03 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2020-10

CONDITIONS: Carcinoma, Renal Cell; Clear Cell Renal Cell Carcinoma
Keywords: clear cell renal cell carcinoma; PET/CT imaging; 89Zr-girentuximab; pharmacokinetics; pharmacodynamics; safety; Diagnostic imaging; 89Zr-TLX250
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: open-label, safety, pharmacokinetic, diagnostic, prospective, multi-center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 89Zr-girentuximab (Experimental): A single administration of 37 Megabecquerel (MBq) (±10%) 89Zr-girentuximab, containing a mass dose of 10 mg of girentuximab
  Interventions: Diagnostic Test: 89Zr-girentuximab

INTERVENTIONS:
Diagnostic Test: 89Zr-girentuximab — A single dose of 37 MBq (±10%) is administered. The dose per dose is equivalent to girentuximab 10 mg (±10%).
  Other Names: 89Zr-TLX250; 89Zr-DFO-TFP-girentuximab (GTX)

SUMMARY:
89Zr-TLX250 is a carbonic anydrase IX (CAIX)-targeted imaging agent that is under clinical development as a non-invasive diagnostic imaging agent for teh detection of clear cell renal cell carcinoma (ccRCC). The Phase 1 study part of this study is to confirm the safety/tolerability and to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) in subjects with suspected renal cell carcinoma (RCC) including clear cell renal cell carcinoma. The Phase 2 component of the study is to to evaluate the sensitivity/specificity of using 89Zr-TLX250 PET/CT images to detect RCC and ccRCC in patients with suspected RCC.

DETAILED DESCRIPTION:
Phase 1:

The phase 1 component of this study will be conducted in in 6-10 subjects at one study center, with the objective of confirming the safety/tolerability and the whole-body dose distribution of 89Zr-TLX250. 89Zr-TLX250 will be administered via a single IV injection (at least 3 min) at an activity dose of 37 MBq (± 10%) and at a dose of 10 mg (±10%). After the enrollment of 6 subjects, if the male-to-female ratio is different from the Japanese epidemiological RCC data (male-to-female ratio ≒ 2:1 in 2017), more subjects, up to 10 subjects in total, are to be enrolled.

Blood sampling for pharmacokinetic analysis will be is performed at 0.5, 1, 2, 4, 24, 72 h and during the Day 5 ± 2 imaging visit. The dose distribution will be determined using low-dose, non-contrast-enhanced CT whole body imaging at 0.5, 4, 24, 72 h and Day 5 ± 2. Diagnostic images will be acquired on Day 3 and Day 5 ± 2 using whole body PET/CT-imaging where individual organs will be assessed using Medical Internal Radiation Dose (MIRD) method.

Seven days after the Day 5 ± 2 imaging visit, patients will attend a follow-up visit to conduct safety evaluations and to undergo blood sampling for HACA measurement.

Phase 2:

The phase 2 component of this study will be conducted after the completion of the phase 1 study in 6-10 patients. This part of the study is equivalent to a phase 2, open-label, multi-center (2-5 sites) to assess the sensitivity/specificity of PET/CT images in subjects with suspected but not definitely diagnosed RCC including ccRCC. The study is intended to evaluate the sensitivity and specificity of PET/CT test as a non-invasive test with the CAIX-targeted imaging agent 89Zr-TLX250. The study will include patients who are scheduled to undergo a partial or total nephrectomy. Patients with an indeterminate renal mass with the longest diameter of 7cm or less, by diagnostic imaging, will receive a single administration of 37 MBq (+/- 10%) 89Zr-TLX250. Imaging will then be conducted Day 5 ± 2 post administration. The partial/total nephrectomy will be performed at institutional discretion any time following the PET/CT imaging visit, but no later than 90 days post administration of 89Zr-TLX250. Histological tumour samples will be prepared and used for histological diagnosis of the renal mass (ccRCC or non-ccRCC) read by a central laboratory.

Image data analyses will be performed by a central image core lab. Qualitative visual analysis (presence or absence of localised 89Zr-TLX250 uptake inside or in vicinity of renal lesion, as seen on contrast-enhanced CT or MRI), will be used to assess test performance or 89Zr-TLX-250 PET/CT imaging to non-invasively detect ccRCC, using histological results from the central histological reference laboratory as standard of truth.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

1. Written and voluntarily given informed consent
2. Aged ≥20 years at the time of enrollment
3. Suspected renal cell carcinoma who have been diagnosed with a renal mass by CT or MRI performed within 90 days before screening
4. Sufficient life expectancy to participate in the study
5. Consent to practice barrier contraception (condoms) until a minimum of 42 days and 90 days after 89Zr-TLX250 administration in female and male, respectively

Phase 2 Part

1. Written and voluntarily given informed consent
2. Aged ≥20 years at the time of enrollment
3. Imaging evidence of a single indeterminate renal mass of ≤ 7 cm in largest diameter on CT or MRI within 90 days prior to screening
4. Scheduled for lesion resection as part of regular diagnostic work-up within 90 days from planned 89Zr-TLX250 administration
5. Sufficient life expectancy to undergo nephrectomy
6. Consent to practice barrier contraception (condoms) until a minimum of 42 days and 90 days after 89Zr-TLX250 administration in female and male, respectively

Exclusion Criteria:

Commonly applied for Phase 1 part and Phase 2 part

1. Those who have hypersensitivity to Girentuximab or DFO
2. Patients with metastatic renal tumor
3. Patients who need treatment for other active malignancies during the study period
4. Patients who have undergone chemotherapy, radiation therapy, or immunotherapy within 4 weeks before the administration of the investigational drug, or have continued adverse events of grade 1 (defined in NCI-CTCAE v5.0) or higher
5. Patients scheduled for anticancer drug treatment during the period from administration of investigational drug to image collection
6. Patients who have been exposed to mouse or chimeric antibody within the past 5 years
7. Patients who have been administered some kind of radionuclide earlier than 10 half-lives of the nuclide.
8. Patients with severe, but not fatal disease, for which the principal investigator / investigator has determined that study participation is not appropriate
9. Women who are pregnant or breastfeeding. And women with childbearing potential who are not pregnant or breastfeeding but suspected of being pregnant by the blood test at screening and pre-dose (within 24 hours before administration). Pre-dose blood pregnancy test can be replaced with urine test
10. Patients who have been administered the drug by any clinical study or clinical trial within 30 days before the scheduled administration of the investigational drug
11. Patients who cannot give legally valid consent by himself / herself
12. Patients with renal dysfunction whose GFR is 60mL / min / 1.73m2 or less
13. Patents who are socially vulnerable (e.g., patients in custody)
14. Others who are judged by the principal investigator or investigator to be inappropriate for participation in this trial Applied only to Phase 2 part 15． Patients whose biopsy is more suitable for pathological diagnosis than partial resection or nephrectomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse events [Safety and Tolerability] | 90 days
  Incidence of abnormal laboratory test results and abnormal vital signs
Determination of the sensitivity and specificity of 89Zr-TLX250 to detect clear cell renal cell carcinoma | 90 days
  The sensitivity and specificity of 89Zr-TLX250 to detect renal cell carcinoma will be established by a diagnostic scan after administration of the investigational product followed by surgery of the indeterminate mass. After surgical removal of the kidney mass , diagnostic histology of the mass will be conducted and used as the "standard of truth" comparator.

SECONDARY OUTCOMES:
Phase 1: Evaluation of the radioactivity distribution and biodistribution/tumor uptake | 0.5, 4, 24, and 72 hours and Day 5 ± 2
  Whole body PET/CT imaging (from the base of skull to the thigh) performed post-injection using non-contrast-enhanced and low-dose CT for absorption correction.
Phase 1: Assessment of tumor uptake | Day 3-5
  This outcome will be evaluated by determining the absorbed dose after injection with 89Zr-TLX250 in identifiable tumor regions taking into account the tumor volume estimated from imaging performed prior to participation to the study.
Phase 2: To evaluate positive predictive value (PPV) of 89Zr-girentuximab PET/CT imaging to detect ccRCC in patients with indeterminate solid renal masses | At end of study , on average of 5 months
  Positive predictive value (PPV) in detecting ccRCC by PT/CT imaging using 89Zr-TLX250 in subjects with undiagnosed solid renal mass
Phase 2: To evaluate negative predictive value (NPV) of 89Zr-girentuximab PET/CT imaging to detect ccRCC in patients with indeterminate solid renal masses | At end of study , on average of 5 months
  Negative predictive value (NPV) using 89Zr-TLX250 in subjects with undiagnosed solid renal mass
To evaluate accuracy of 89Zr-girentuximab PET/CT imaging to detect ccRCC in patients with indeterminate solid renal masses | At end of study , on average of 5 months
  Determine accuracy in detecting ccRCC by PT/CT imaging using 89Zr-TLX250 in subjects with undiagnosed solid renal mass
Phase 2: To evaluate the correlation between 89Zr- girentuximab SUVs and degree of histological carbonic anhydrase IX (CAIX) expression | Within 90 days
  This outcome will be assessed on all patients. The counts derived from the PET/CT imaging of the renal lesion will be compared with the amount of CAIX expressed in the histologically extracted sample
Phase 2: To evaluate inter-reader variability of diagnostic assessments of 89Zr- girentuximab PET/CT images, when performed by multiple readers | This analysis will be conducted through study completion, on average of 5 months
  This outcome will be conducted on all patients. Three blinded readers operating independently will be used to read each patient PET/CT image and determine if the target lesion is positive for Zr89. A comparison of findings will then be made between the readers for each patient individually.
Phase 2: Assessment of differences in a same reader | This analysis will be conducted through study completion, on average of 5 months
  The difference in evaluations of 89Zr-TLX250 PET/CT images by a same reader is assessed with the use of Cohen's κ coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Noboru Nakaigawa, MD, PhD, Principal Investigator — Yokohama City University Hospital
Locations (1):
- Yokohama City University Hospital, Yokohama, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No